CLINICAL TRIAL: NCT04886752
Title: The Effect of Liposome Vitamin C on the Absorption
Brief Title: The Effect of Liposome Vitamin C on the Absorption and Metabolism of the Human Body.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201903113RSA
Record Dates: First submitted 2021-05-09; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Vitamin C Deficiency
MeSH Terms: conditions — Ascorbic Acid Deficiency | interventions — Ascorbic Acid; Liposomes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin C without liposome (Sham Comparator): vitamin C without liposome
  Interventions: Dietary Supplement: vitamin C without liposome
- liposomal process A vitamin C (Placebo Comparator): liposomal process A vitamin C
  Interventions: Dietary Supplement: liposomal process A vitamin C
- liposomal process B vitamin C (Double Nutri™) (Experimental): liposomal process B vitamin C (Double Nutri™)
  Interventions: Dietary Supplement: liposomal process B vitamin C (Double Nutri™)

INTERVENTIONS:
Dietary Supplement: vitamin C without liposome — subjects need to take 3 tests during trail. After each test was completed, a washout period of 14 days was required before the next test start
  Arms: vitamin C without liposome
Dietary Supplement: liposomal process A vitamin C — subjects need to take 3 tests during trail. After each test was completed, a washout period of 14 days was required before the next test start
  Arms: liposomal process A vitamin C
Dietary Supplement: liposomal process B vitamin C (Double Nutri™) — subjects need to take 3 tests during trail. After each test was completed, a washout period of 14 days was required before the next test start
  Arms: liposomal process B vitamin C (Double Nutri™)

SUMMARY:
To evaluate the difference between vitamin C in the form of oral liposomes and general vitamin C in a fixed period of time in plasma and urine.

DETAILED DESCRIPTION:
we recruited 11 healthy subjects and adopted a cross-over test. the subjects need to take 3 tests during trail. After each test was completed, a washout period of 14 days was required before the next test start. The subjects were informed to consume one sachet vitamin C without liposome, liposomal process A vitamin C, or liposomal process B vitamin C (Double Nutri™) every test, and vitamin C concentration was measured at baseline (0 hours), 0.5, 1, 2, 3, 4, and 8 hours after taking test sample.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 20-60 years old,
2. No heart, liver, kidney, endocrine and major organic diseases

Exclusion Criteria:

1. Renal insufficiency and dialysis
2. Cancer
3. Underweight (BMI≦17) or obese (BMI≧27),
4. Take chronic disease drugs,
5. Blood pressure systolic blood pressure ≧130 mmHg or diastolic blood pressure ≧85 mmHg,
6. Too high fasting blood glucose ≧ 100 mg/dL,
7. Triglyceride ≧ 150 mg/dL,Total cholesterol ≧ 200 mg/dL,
8. Have a history of vitamin C allergy,
9. People with mental illness,
10. Pregnant or breastfeeding women,
11. Hematosis,
12. Kidney stones,
13. Long-term vitamin C supplements (at least 200 mg per day for more than one month)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
vitamin c detection | at 8 hours after taking test sample
  vitamin c was assessed by Ascorbic Acid Colorimetric Assay Kit II
The change of Triglyceride | at 8 hours after taking test sample
  Venous blood was sampled to measure concentrations of Triglyceride
The change of body mass index (BMI) | Time 0, 0.5, 1, 2, 3, 4, and 8 hours after taking test sample
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass.The body mass index (BMI, kg/m^2) and body mass (kg) were assessed by InBody770.
The change of aspartate aminotransferase | at 8 hours after taking test sample
  Venous blood was sampled to measure concentrations of aspartate aminotransferase
The change of alanine aminotransferase | at 8 hours after taking test sample
  Venous blood was sampled to measure concentrations of alanine aminotransferase
The change of creatine | at 8 hours after taking test sample
  Venous blood was sampled to measure concentrations of creatine

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Shiun Tsai, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Research & Design Center, TCI CO., Ltd, Taipei, Taiwan